CLINICAL TRIAL: NCT04138485
Title: A Randomized, Multicenter, Double-Blind, Placebo Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of IgPro10 (Intravenous Immunoglobulin, Privigen®) for the Treatment of Adults With Systemic Sclerosis
Brief Title: Efficacy and Safety of IgPro10 in Adults With Systemic Sclerosis (SSc)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to business reasons, not safety issues
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IgPro10_2001; 2019-000906-31 (EudraCT Number)
Record Dates: First submitted 2019-10-14; First posted 2019-10-24 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — gamma-Globulins; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IgPro10 (Experimental): 10% liquid formulation of human immunoglobulin for intravenous use
  Interventions: Biological: IgPro10
- Placebo (Placebo Comparator): 0.5% human albumin solution stabilized with 250 mmol/L L-proline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: IgPro10 — 10% liquid formulation of human immunoglobulin for IVIG
  Other Names: Human normal immunoglobulin
  Arms: IgPro10
Biological: Placebo — 0.5% human albumin solution stabilized with 250 mmol/L L-proline
  Other Names: Albumin
  Arms: Placebo

SUMMARY:
This randomized, multicenter, double-blind (DB), placebo controlled, phase 2 study will evaluate the efficacy and safety of IgPro10. The DB Treatment Period will be followed by a 24-week Open-label (OL) Treatment Period.

Eligible subjects will be randomized at Baseline in a 2:1 ratio of treatment IgPro10 or placebo in the DB Treatment Period. All subjects who enter OL Treatment Period will receive IgPro10.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years (male or female) at time of providing written informed consent
* Documented diagnosis of SSc according to ACR / EULAR criteria 2013
* mRSS ≥ 15 and ≤ 45
* Disease duration ≤ 5 years defined as the time from the first non-Raynaud's phenomenon manifestation
* Subjects within first 18 months of disease duration from first non-Raynaud's phenomenon manifestation.

Exclusion Criteria:

* Primary rheumatic autoimmune disease other than dcSSc, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, mixed connective tissue disorder, polymyositis, and dermatomyositis, as determined by the investigator Note: Subjects with fibromyalgia, secondary Sjogren's syndrome, and scleroderma-associated myopathy or myositis at Screening are not excluded
* Positive anti-centromere autoantibodies at Screening
* Evidence of severe chronic kidney disease with estimated glomerular filtration rate < 45 mL/min/1.73 m2 (as calculated by the Chronic Kidney Disease Epidemiology Collaboration equation) or receiving dialysis. Additionally, subjects with current confirmed diagnosis of diabetes mellitus and requiring medication, with eGFR < 90 mL/min/1.73m2 will be excluded from the study.
* History of documented thrombotic episode eg, PE, DVT, myocardial infarction, thromboembolic stroke at any time Note: past superficial thrombophlebitis more than two years from Screening is not exclusionary
* Documented thrombophilic abnormalities including blood hyperviscosity, protein S or protein C deficiency, anti-thrombin-3 deficiency, plasminogen deficiency, antiphospholipid syndrome, Factor V Leiden mutation, dysfibrinogenemia, or prothrombin G20210A mutation
* Greater than 3 specified current risk factors for TEEs (documented and currents conditions): atrial fibrillation, coronary disease, diabetes mellitus, dyslipidemia, hypertension, obesity (Body Mass Index ≥ 30 kg/m2), recent significant trauma, and immobility (wheelchair-bound or bedridden)
* Ongoing active serious infection at Screening (including, but not limited to, pneumonia, bacteremia/septicemia, osteomyelitis/septic arthritis, bacterial meningitis, or visceral abscess)
* Malignancy in the past 2 years, except for non-melanoma skin cancer, cervical carcinoma in situ, or other in situ cancer if it has been excised and treated within in the past year
* Known hypoalbuminemia, protein-losing enteropathies, and any proteinuria (defined by total urine protein concentration > 0.2 g/L)
* Known IgA deficiency or serum IgA level < 5% lower limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Response on American College of Rheumatology Combined Response Index in Diffuse Systemic Sclerosis (ACR CRISS) score in IgPro10 vs Placebo | Over 48 weeks

SECONDARY OUTCOMES:
Proportion of subjects meeting cardiopulmonary or renal failure criteria in ACR CRISS Step 1 events | Over 48 weeks
Proportion of responders (ACR CRISS > 0.6) | Over 48 weeks
Mean change from Baseline in Modified Rodnan Skin Score (mRSS) | Baseline and over48 weeks
Mean change from Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) | Baseline and over 48 weeks
Mean change from Baseline in Forced Vital Capacity (FVC)% predicted | Baseline and over 48 weeks
Mean change from Baseline in diffusing capacity of lung for carbon monoxide (DLCO)% predicted | Baseline and over 48 weeks
Mean change from Baseline in Physician Global Assessment (MDGA) | Baseline and over 48 weeks
  MDGA evaluates the overall impact of SSc on the participant as assessed by the physician on a 11-point Numeric rating scale scale from 0 (excellent) to 10 (extremely poor)
Mean change from Baseline in Patient Global Assessment (PGA) | Baseline and over 48 weeks
  PGA evaluates the overall impact of SSc on the participant as assessed by the physician on a 11-point Numeric rating scale scale from 0 (excellent) to 10 (extremely poor)
Mean change from Baseline in UCLA Scleroderma Clinical Trial Consortium Gastrointestinal Tract 2.0 (UCLA SCTC GIT 2.0) total score and subscale | Baseline and over 48 weeks
  This survey consists of 34 questions and items are scored on a scale of 0 (better health) to 3 (worse health). Scores are combined to form total score.
Mean change from Baseline in Scleroderma Skin Patient Reported Outcome (SSPRO) score in IgPro10 vs Placebo | Baseline and up to 48 weeks
Proportion of responders in mRSS | Up to 48 weeks
  Response is decrease of mRSS ≥ 5 points and change of ≥ 25% from Baseline in IgPro10 vs Placebo
Time to treatment failure (time from first infusion to time of first event) in IgPro10 vs Placebo | Over 48 weeks
  Treatment failure - defined as occurrence of SSc associated complications in ACR CRISS step 1 events, digital ischemia (requiring hospitalization for IV prostacyclin, surgical intervention or amputation), serious gastrointestinal events (events requiring parenteral nutrition due to SSc -such as total parenteral nutrition or enteral nutrition), all-cause mortality
Proportion of subjects with events at Week 48 in IgPro10 vs Placebo | Over 48 weeks
  Events defined as occurrence of SSc associated complications in ACR CRISS step 1 events, digital ischemia (requiring hospitalization for IV prostacyclin, surgical intervention or amputation), serious gastrointestinal events (events requiring parenteral nutrition due to SSc -such as total parenteral nutrition or enteral nutrition), all -cause mortality
Mean change from Baseline in Cochin Hand Function Scale in IgPro10 vs Placebo | Baseline and over 48 weeks
Mean change from Baseline in Scleroderma Health Assessment Questionnaire (SHAQ) score in IgPro10 vs Placebo | Baseline and over 48 weeks
Mean change from baseline in muscle strength as measured by Manual Muscle Testing 8 (MMT) in IgPro10 vs Placebo | Baseline and over 48 weeks
Number of subjects with adverse events (AEs) including any AEs, treatment-emergent AEs (TEAEs), serious AEs (SAEs), and AEs of special interest (AESIs) | Over 48 weeks
Percentage of subjects with AEs, TEAEs, SAEs, AESIs | Over 48 weeks
Concentration of serum trough IgG levels at Baseline and prior to first infusion | Baseline and up to 72 weeks
Mean change from Baseline in Modified Rodnan skin score (mRSS) | Baseline and over 72 weeks
Mean change from Baseline in Patient global assessment (PGA) | Baseline and over 72 weeks
Proportion of responders (ACR CRISS > 0.6) | Over 72 weeks
Mean change from Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) | Baseline and over 72 weeks
Mean change from Baseline in Forced Vital Capacity (FVC)% predicted | Baseline and over 72 weeks
Mean change from Baseline in diffusing capacity of lung for carbon monoxide (DLCO)% predicted | Baseline and over 72 weeks
Mean change from Baseline in Physician Global Assessment (MDGA) | Baseline and over 72 weeks
Number of subjects with adverse events (AEs) including any AEs, treatment-emergent AEs (TEAEs), serious AEs (SAEs), and AEs of special interest (AESIs) | Over 72 weeks
Percentage of subjects with AEs, TEAEs, SAEs, AESIs | Over 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (77):
- United States (20):
  - Mayo Clinic Arizona - Scottsdale, Scottsdale, Arizona
  - Pacific Arthritis Care Center, Los Angeles, California
  - University of California, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Lombardi Cancer Center-Georgetown University, Washington D.C., District of Columbia
  - Alliance for Multispecialty Research, Wichita, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - John Hopkins Bayview Medical Center, Baltimore, Maryland
  - Boston University Amyloidosis Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Rutgers Clinical Research Center, New Brunswick, New Jersey
  - Northwell Health, Great Neck, New York
  - Hospital For Special Surgery, New York, New York
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - Altoona Center For Research, Duncansville, Pennsylvania
  - University of Pennsylvania - Perelman Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University Of Texas Medical School At Houston (Utms), Houston, Texas
- Argentina (4):
  - APRILLUS Asistencia e Investigacion Clinica, Buenos Aires
  - Hospital Militar Central, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Sanatorio Parque S.A y Consultorios Externos Asociados, Rosario
- Australia (2):
  - John Hunter Hospital / Autoimmune Resource and Research Centre, New Lambton Heights, New South Wales
  - PARC Clinical Research, Adelaide, South Australia
- Belgium (2):
  - UZ Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Mount Sinai Hospital, The Rebecca Macdonald Centre For Arthritis, Toronto, Canada
- France (7):
  - CHU de Caen, Caen
  - CHRU de Lille Hopital Huriez, Lille
  - Internal Medicine, Nantes University Hospital, Nantes
  - Assistance Publique - Hopitaux de Paris (AP-HP), Paris
  - CHU de Rennes-Hopital Sud, Rennes
  - Centre Hospitalier Universitaire de Rouen-Hopital, Rouen
  - CHU Hautepierre, Strasbourg
- Germany (9):
  - Kerckhoff Klinik GmbH, Abteilung für Rheumatologie und Klinische Immunologie Rheumatologie, Bad Nauheim
  - Charite - Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin
  - University Hospital of Cologne, Cologne
  - Universitaetsklinikum Freiburg- Klinik fuer Rheumatologie und Klinische Immunologie, Freiburg im Breisgau
  - Universitaetsmedizin der Johannes Gutenberg, Mainz
  - University Hospital Of Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - Hospital St. Josef, Wuppertal
- Italy (10):
  - Universita degli Study di Ancona, Ancona
  - Universita Degli Studi Di Bari Aldo Moro, Bari
  - Universita degli Studi Di Brescia, Brescia
  - Universita degli Studi Firenze, Florence
  - UOC Immunoreumatologia, L’Aquila
  - Azienda Ospedaliera Gaetano Pini, Milan
  - Modena University, Modena
  - Universita degli Studi di Napoli Federico II, Napoli
  - IRCCS Policlinico San Matteo, Pavia
  - Dip.to Med. Sperimentale -Polic.Umberto I -Univ. La Sapienza, Rome
- Mexico (6):
  - Centro Integral en Reumatologia, SA de CV, Guadalajara
  - Centro De Estudios De Investigation Basica Y Clinica S.C, Jalisco
  - Cliditer, S.A. DE C.V., Mexico City
  - Centro de Investigacion y Tratamiento Reumatologico S.C., Mexico City
  - Instituto Nacional De Ciencias Medicas Y Nutricion, México
  - Centro de Alta Especialidad en Reumatologia, San Luis Potosí City
- Poland (5):
  - Uniwersytecki Szpital Kliniczny W Bialymstoku, Bialystok
  - University Clinical Centre, Medical University of Gdansk, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny, Katowice
  - Klinika Dermatologii Szpital im. Dzieciątka Jezus, Warsaw
  - Klinika i Poliklinika Układowych Chorób Tkanki Łącznej Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji, Warsaw
- Spain (7):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Universitari Materno Infantil Vall Dhebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Univ 12 de Octubre, Madrid
  - Hospital Infanta Luisa Quirónsalud, Seville
  - Hospital Universitari Dr.Peset, Valencia
- Cantonal Hospital St. Gallen - Klinik fuer Rheumatologie, Sankt Gallen, Switzerland
- United Kingdom (3):
  - Countess of Chester Hospital, Chester
  - Chapel Allerton Hospital, Leeds
  - Royal Free Hospital-Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systemic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.